CLINICAL TRIAL: NCT06146023
Title: Preclinical Performance of The Combined Application of Two Robotic Systems in Microsurgery
Brief Title: Performance of Robotic Microsurgery Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Kai Wessel, Principal Investigator, University Hospital Muenster
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000034951
Record Dates: First submitted 2023-11-10; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Robotic Surgery; Microsurgery; Anastomosis
Keywords: Learning curve; Robotics; Surgical ergonomics; Surgical training

STUDY DESIGN:
Intervention Model Description: Comparison of conventional manual microsurgery versus robot-assisted microsurgery
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded for participant groups and number of anastomosis during evaluation of scores.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Conventional (Active Comparator): Conventional microsurgery with conventional microsurgical instruments and conventional surgical microscope
  Interventions: Procedure: Conventional anastomosis
- Robotic (Experimental): Robot-assisted microsurgery with microsurgery robot and robotic microscope
  Interventions: Device: Robotic anastomosis (Symani surgical system and RoboticScope)

INTERVENTIONS:
Device: Robotic anastomosis (Symani surgical system and RoboticScope) — Robot-assisted microvascular anastomosis on 1.0-mm-diameter silicone vessels using the Symani surgical system and RoboticScope
  Arms: Robotic
Procedure: Conventional anastomosis — Conventional microvascular anastomosis on 1.0-mm-diameter silicone vessels using conventional microsurgical instruments and conventional surgical microscope
  Arms: Conventional

SUMMARY:
The goal of this preclinical trial is to learn about the benefits and limitations of novel robotic devices for microsurgery, based on different levels of microsurgical experience. The main questions it aims to answer are:

Is robot-assisted microsurgery faster, better and more ergonomic than conventional microsurgery in a preclinical standardized setting?

Participants will perform microvascular anastomoses on 1.0-mm-diameter artificial silicone vessels using a conventional manual approach versus a novel robot-assisted approach. Researchers will compare the performance of novices, advanced participants and experts to evaluate the role of microsurgical experience when learning the new technique.

DETAILED DESCRIPTION:
Recent advancements in the development of robotic devices increasingly draw the attention towards the concept of robotic microsurgery, as several systems tailored to open microsurgery are being introduced. This study describes the combined application of a novel microsurgical robot, the Symani, with a novel robotic microscope, the RoboticScope, for the performance of microvascular anastomoses in a two-center preclinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Novices: no prior experience in microsurgery
* Residents: 2-4 years of experience in microsurgery
* Experts: at least 5 years of experience in microsurgery

Exclusion Criteria:

* previous training with the robotic devices applied in this study
* contraindications for usage of robotic devices (magnetic field)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Surgical time | Duration of anastomosis
  Time to perform anastomosis in minutes and seconds.
Anastomosis quality | Evaluated right after completion of each anastomosis
  Anastomosis lapse index (ALI) to evaluate the quality of each stitch. Score indicates absolute number of errors per anastomosis. Low values indicate better results.
Microsurgical skills | Duration of anastomosis
  Structured assessment of microsurgery skills (SAMS) to evaluate microsurgical skill acquisition. Score includes 8 items evaluated from 1 (minimum) to 5 (maximum). High values indicate better results.

SECONDARY OUTCOMES:
Subjective Satisfaction | Evaluated right after completion of each anastomosis
  Satisfaction with anastomosis und robotic performance (Questionnaire). Evaluation of anastomosis and robotic devices from 1 (minimum) to 10 (maximum). High values indicate better results.
Surgical ergonomics | Evaluated right after completion of each anastomosis
  Rapid entire body assessment (REBA) to evaluate surgical ergonomics. Numeric score, low values indicate better results.

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Kückelhaus, MD, Principal Investigator — University Hospital Muenster; Haripriya S Ayyala, MD, Principal Investigator — Yale University
Locations (2):
- Yale New Haven Hospital, New Haven, Connecticut, United States
- University Hospital Muenster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No
Primary data from this study can be made available upon request for dedicated purposes.